CLINICAL TRIAL: NCT05362838
Title: Conventional Laparoscopy Versus Robotic Surgery for Pain Relief in Patients With Deep Infiltrating Endometriosis: a Pilot Study.
Brief Title: Conventional Laparoscopy Versus Robotic Surgery for Pain Relief in Patients With Deep Infiltrating Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christine Bekos, Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIE pain robotic vs. LSK
Record Dates: First submitted 2022-05-03; First posted 2022-05-05 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Endometriosis; Endometriosis-related Pain; Endometriosis Pelvic
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robotic-assisted laparoscopy (Active Comparator): The robotic-assisted resection of endometriosis will be performed using the da Vinci Surgical System Si (Intuitive Surgical) using up to five ports as needed. An umbilical port will be placed for the laparoscope (10/12 mm), a 5-mm port for the assistant, and two to three ports (5/8 mm) for the robotic arms.
  Interventions: Procedure: robotic-assisted laparoscopy
- conventional laparoscopy (Active Comparator): Laparoscopic-assisted cystectomy of endometrioma will be performed using up to four 5-mm ports, including an umbilical port and additional ports as dictated by each individual surgery.
  Interventions: Procedure: Conventional laparoscopy

INTERVENTIONS:
Procedure: robotic-assisted laparoscopy — Superficial and deep endometriosis resection will be performed in the usual standard fashion. All superficial lesions suspicious for endometriosis (pigmented and nonpigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy will be performed for endometriomas. Additional procedures are performed as needed to completely resect all endometriosis lesions. The fascia of any port ≥10 mm will be reapproximated. If bowel resection and re-anastomosis is necessary this will be performed together with a General Surgeon.
  Other Names: DaVinci laparoscopy
  Arms: robotic-assisted laparoscopy
Procedure: Conventional laparoscopy — Superficial and deep endometriosis resection will be performed in the usual standard fashion. All superficial lesions suspicious for endometriosis (pigmented and nonpigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy will be performed for endometriomas. Additional procedures are performed as needed to completely resect all endometriosis lesions. The fascia of any port ≥10 mm will be reapproximated. If bowel resection and re-anastomosis is necessary this will be performed together with a General Surgeon.
  Arms: conventional laparoscopy

SUMMARY:
Background: Endometriosis is a common disease, affecting women in their reproductive age suffering from infertility, adnexal masses and chronic pelvic pain, obstruction of the bowel or urinary tract. Deeply infiltrating endometriosis (DIE) is defined as a solid endometriosis mass situated more than 5 mm deep to the peritoneum. These lesions are considered very active and are strongly associated with pelvic pain symptoms.

Surgery is recommended in women with pain resistant to medical therapy and in women with contraindications to or refusal of medical therapy. Further indications for surgical treatment are the need of excluding malignancy in an adnexal mass, obstruction of the bowel or urinary tract. It is hypothesized that in patients with lesions in complex anatomic sites, a robot-assisted approach may provide improved instrument articulation compared with conventional laparoscopy, but no data are available.

Aims: The aim of this study is to perform a pilot study investigating differences between robot-assisted laparoscopy compared to conventional laparoscopy regarding subjective symptom outcome, evaluated by VAS score for non-menstrual pelvic pain and dysmenorrhea.

Study population: The study population will consist of women aged between 18 and 51 years who are referred to our gynecologic outpatient clinic due to symptomatic endometriosis. Women with suggested DIE and an indication for surgery can be included in this trial.

Methods: Laparoscopic-assisted resection of endometriosis will be performed using up to five 5-mm ports, including an umbilical port and additional ports as dictated by each individual surgery. The robotic-assisted resection of endometriosis will be performed using the da Vinci Surgical System Si (Intuitive Surgical) using up to five ports as needed. Superficial and deep endometriosis resection will be performed in the usual standard fashion. Histological confirmation of endometriosis will be performed. The primary outcome is subjective symptom improvement. This will be evaluated by visual analog scale (VAS) for dysmenorrhea and non-menstrual pelvic pain on a daily basis for at least 1 calendar month before the operation to obtain adequate baseline measurements. This evaluation will be repeated 3 and 6 months after surgery.

DETAILED DESCRIPTION:
Experimental Plan Study design

This trial is a single-center, prospective, pilot study conducted with the aim of determining differences of robotic surgery compared to simple laparoscopic surgery with regard to the primary outcome in patients with suspected endometriosis. Postoperative follow-up will take place after 3 and 6 months. All women referred to our department for deep endometriosis will undergo clinical examination by a senior surgeon experienced in endometriosis as well as MRI examination. We will include all patients with suspected DIE affecting Enzian compartments A, B and C with lesions sized ≥1 (A2-3, B2-3 and C2-3). In cases with colorectal involvement, irrigoscopy will be used to check for digestive tract stenosis and associated digestive tract localizations. Complementary examinations, such as cystoscopy will be performed in women with associated involvement of urinary tract.

In women with pregnancy intention and deep endometriosis, an exhaustive assessment of the disease will systematically be performed before deciding between primary surgery and primary assisted reproductive techniques.

Gynecological examination is performed at each visit. Furthermore, subjective outcome will be assessed with standardized questionnaires.

Study setting Participants and recruitment The study population will consist of women aged between 18 and 51 years who are referred to our gynecologic outpatient clinic due to symptomatic endometriosis. Women with suggested DIE affecting Enzian compartments A, B and C with lesions sized ≥1 (A2-3, B2-3 and C2-3) and an indication for surgery can be included in this trial.

Intervention Laparoscopic-assisted resection of endometriosis will be performed using up to four 5-mm ports, including an umbilical port and additional ports as dictated by each individual surgery. The robotic-assisted resection of endometriosis will be performed using the da Vinci Surgical System Si (Intuitive Surgical) using up to five ports as needed. An umbilical port was placed for the laparoscope (10/12 mm), a 5-mm port for the assistant, and two or three ports (5/8 mm) for the robotic arms. Superficial and deep endometriosis resection will be performed in the usual standard fashion. All lesions suspicious for endometriosis (pigmented and nonpigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect. Cystectomy will be performed for endometrioma(s). Additional procedures are performed as needed to completely resect all endometriosis lesions. The fascia of any port ≥10 mm will be reapproximated. If bowel resection and re-anastomosis is necessary this will be performed together with a General Surgeon.

Participating surgeons will be defined as high volume surgeons in endometriosis surgery and will also be part of the endometriosis core team.

Histological confirmation of endometriosis will be performed.

Postoperative Management: The patients are instructed to rest for 2 weeks after the operation (not to work, to do sport, to do the cleaning and to carry more than five kilos). They are allowed to return to work after 2 weeks and to take part in sport or have intercourse after 6 weeks. Follow-up visits are scheduled after 3 and 6 months in our outpatient clinic due to our study protocol.

Inclusion and exclusion criteria In the present study, we will include women with suspected deep infiltrating endometriosis. The disease will be classified according to the ENZIAN score by the surgeon.

Inclusion criteria

* Suspected deep infiltrating endometriosis affecting Enzian compartments A, B and C with lesions sized ≥1 (A2-3, B2-3 and C2-3)
* Mean VAS score for dysmenorrhea or non-menstrual pelvic pain >= 5 (assessed at 5 days/ month with the heaviest symptoms)
* Surgical endometriosis resection is planned

Exclusion criteria

* History of malignant diseases
* Current systemic glucocorticoid or immunosuppressant treatment
* Subject is unable or unwilling to participate
* Postmenopausal women
* Combined oral contraception

Data collection At baseline, the following data will be collected: demographics and medical history data (age, body mass index, parity, menopausal and hormone therapy status, current smoking, previous operations, and medical comorbidities (diabetes mellitus, connective tissue disorders)). Previous endometriosis-specific treatments and responses will be assessed. Patients will be asked to complete the Patient Global Impression of Change (PGIC) and the Endometriosis Health Profile (EHP) EHP-30. Gynecological examination is performed at each visit.

The patients will be asked to rate their satisfaction with the appearance of their scars on a 10-point Likert scale (with 1 being very unsatisfied and 10 being very satisfied). Similar scales have been used successfully in previous trials assessing satisfaction with scars.

Postoperative follow up visits will be performed after 3 and 6 months following the operation.

Primary and secondary outcome measures The primary outcome is subjective symptom improvement. This will be evaluated by Visual analog scale (VAS) for dysmenorrhea and non-menstrual pelvic pain on a daily basis for at least 1 calendar month before the operation to obtain adequate baseline measurements. This evaluation will be repeated 3 and 6 months after surgery. In detail, this means that patients will be asked to complete a VAS for dysmenorrhea and non-menstrual pelvic pain on a daily basis for at least 1 calendar month after 3 months and after 6 months following the operation. For VAS score we will calculate the mean of the 5 days/months with the highest VAS score. PGIC will be used to calculate the rate of responders.

Next to pain, medication being taken for endometriosis-associated pain and menstrual bleeding will be assessed in this daily questionnaire. Patients will be asked to write down their VAS score before taking pain medication.

The secondary outcomes are the Biberoglu and Behrman (B&B) score, the rate of adverse events related to surgery both intraoperative (bladder injury, bowel injury, ureteral obstruction, massive bleeding) but also postoperative (classified using Clavien Dindo classification), operation time, length of hospitalization, blood loss (change of hemoglobin levels 24 hours after surgery), laparotomic conversion rate and use of pain killers during the hospital stay.

Dyspareunia, bladder pain, dyschezia, fatigue and abnormal vaginal bleeding will be assessed.

Patients will be asked to finish three questionnaires: the Patient Global Impression of Change 14, the Endometriosis Health Profile (EHP) EHP-30 and a 10-point Likert scale for cosmetic satisfaction.

Disease recurrence rate up to 12 months after surgery will be assessed. Endometriosis recurrence can have different levels: symptoms recurrence based on patient history (VAS pain score ≥ 5), but no proof of recurrence by imaging and/or surgery; endometriosis recurrence based on non-invasive imaging in patients with or without symptoms; recurrence of histologically proven endometriosis: when the patient is re-operated, endometriosis is visually observed and confirmed histologically.

Sample size and power considerations Due to missing results for pain assessment comparing patients with endometriosis after conventional laparoscopy versus robotic surgery a pilot study including 50 (25 versus 25) patients in total will be performed. The distribution to both groups will be performed randomly using a computer-based randomizer. Stratification for VAS score (5-7 versus 8-10) and the surgeon will be performed. The results from this pilot study will be the basis for future randomized-controlled studies.

The pre-post-OP changes in VAS-Score will be compared between 2 different groups: conventional laparoscopy versus robotic surgery. To investigate the difference between groups, one-sided two-sample test of mean changes will be conducted.

Statistical analysis will be performed using SPSS and Excel software. Data will be calculated and graphed as mean plus minus standard error of mean (SEM).

Metric variables will be reported by mean and standard deviation resp. median and IQR, categorical variables will be reported by frequencies per group and timepoint. The primary outcome subjective symptom improvement after 6 months in either group will be analyzed by a t-test or a Man-Whitney-U-test depending on the distribution of improvements.

For the secondary endpoints, changes in B&B score, differences of rates of adverse events between the two treatment groups will be analyzed by a Chi-squared test. Blood loss, use of pain killers and changes in condition-specific quality of life will be compared between groups analogously to the primary outcome.

Statistical significance will be set 0.05. No correction for multiple testing is performed because only one main hypothesis is considered.

ELIGIBILITY:
Inclusion Criteria:

* Suspected deep infiltrating endometriosis affecting Enzian compartments A, B and C with lesions sized ≥1 (A2-3, B2-3 and C2-3)
* Mean VAS score for dysmenorrhea or non-menstrual pelvic pain >= 5 (assessed at 5 days/ month with the heaviest symptoms)
* Surgical endometriosis resection is planned

Exclusion Criteria:

* History of malignant diseases
* Current systemic glucocorticoid or immunosuppressant treatment
* Subject is unable or unwilling to participate
* Postmenopausal women
* Combined oral contraception

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Visual analog scale (VAS) from baseline to 3 and 6 months after the operation | 6 months after the operation
  Patients will be asked to complete a VAS for dysmenorrhea and non-menstrual pelvic pain on a daily basis for at least 1 calendar month at baseline and after 3 months and after 6 months following the operation. For VAS score we will calculate the mean of the 5 days/months with the highest VAS score. Patients will be asked to write down their VAS score before taking pain medication.
Pain medication | 6 months after the operation
  Medication being taken for endometriosis-associated pain will be assessed in this daily questionnaire (type of medication and dosage).
Menstrual bleeding | 6 months after the operation
  Menstrual bleeding will be assessed in this daily questionnaire (yes versus no).
Patients' Global Impression of Change (PGIC) | 6 months after the operation
  PGIC will be used to calculate the rate of responders 3 and 6 months after the operation

SECONDARY OUTCOMES:
Change in Biberoglu and Behrman (B&B) score from baseline to 3 and 6 months after the operation | 6 months after the operation
  postoperative B&B score (3 and 6 months after the operation) compared to preoperative B&B score
rate of intraoperative adverse events | 1 day
  rate of intraoperative adverse events (bladder injury, bowel injury, ureteral obstruction, massive bleeding)
rate of postoperative adverse events | 4 weeks
  rate of postoperative adverse events related to surgery (classified using Clavien Dindo classification)
operation time | 1 day
  operation time in minutes
length of hospitalization (following the operation) | 2 weeks
  length of hospitalization in days
blood loss | 1 day
  change of hemoglobin levels 24 hours after surgery
laparotomic conversion rate | 1 day
  laparotomic conversion rate
change of the Endometriosis Health Profile (EHP) EHP-30 from baseline to 3 and 6 months after the operation | 6 months after the operation
  questionnaires: the Endometriosis Health Profile (EHP) EHP-30 (preoperative versus 3 and 6 months after the operation)
10-point Likert scale for cosmetic satisfaction | 6 months after the operation
  questionnaires: 10-point Likert scale for cosmetic satisfaction 3 and 6 months after the operation
Disease recurrence rate up to 12 months after surgery | 12 months after the operation
  Endometriosis recurrence can have different levels: symptoms recurrence based on patient history (VAS pain score ≥ 5), but no proof of recurrence by imaging and/or surgery; endometriosis recurrence based on non-invasive imaging in patients with or without symptoms; recurrence of histologically proven endometriosis: when the patient is re-operated, endometriosis is visually observed and confirmed histologically.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Wenzl, Prof, Study Director — Medical University of Vienna, Department of Obstetrics and Gynecology
Locations (1):
- Medical University of Vienna, Department of Obstetrics and Gynecology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No